CLINICAL TRIAL: NCT01706627
Title: Melatonin In Cancer Patients Receiving Chemotherapy: A Randomized, Double Blind, Placebo, Controlled Trial
Brief Title: Melatonin In Reduction of Chemotherapy-Induced Toxicity (MIRCIT) Trial
Acronym: MIRCIT
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Khon Kaen University (Other)
Collaborators: Srinagarind Hospital, Khon Kaen University (Other); Khon Kaen Hospital, Khon Kaen (Unknown); General Drugs House Co.,LTD. (Other); Thailand Research Fund (Other)
Responsible Party: Principal Investigator, Nutjaree Pratheepawanit Johns, Associate Professor, Khon Kaen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MIRCIT; TRF (Other Grant/Funding Number: Thailand Research Fund)
Record Dates: First submitted 2012-10-11; First posted 2012-10-15 (Estimated); Last update posted 2012-10-15 (Estimated); Status verified 2012-10

CONDITIONS: Advanced Stage Cancer
Keywords: cancer; melatonin; adjuvant therapy; quality of life; survival; adverse events; oxidative stress
MeSH Terms: conditions — Neoplasms | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Matched placebo (Placebo Comparator): Matched placebo (identical formulation and delivery, without active ingredient)
  Interventions: Drug: Matched placebo
- Drug: 10 mg Melatonin (Active Comparator): 10 mg melatonin gelatin capsule
  Interventions: Drug: 10 mg Melatonin
- Drug: 20 mg Melatonin (Active Comparator): 20 mg melatonin gelatin capsule
  Interventions: Drug: 20 mg Melatonin

INTERVENTIONS:
Drug: 10 mg Melatonin — Active Comparator: Drug: Melatonin 10 mg
  Arms: Drug: 10 mg Melatonin
Drug: 20 mg Melatonin — Active Comparator: Drug: Melatonin 20 mg
  Arms: Drug: 20 mg Melatonin
Drug: Matched placebo — Matched placebo (identical formulation and delivery, without active ingredient)
  Arms: Matched placebo

SUMMARY:
Meta-analysis of previous studies have shown that melatonin is a beneficial adjutant for reducing chemotherapy-induced toxicity; however no randomized, double-blind, placebo controlled trials have been conducted. This study evaluates the effect of melatonin in improving quality of life and reducing chemotherapy-induced toxicity in advanced cancer patients. This is a multi-center, randomized, double-blind, placebo controlled trial conducted in patients with histologically proven advanced non small cell lung, breast, head and neck or sarcoma cancer. Mixed-block randomization, stratified by center and treatment scheme is used to divide eligible patients into three groups: melatonin 20 mg, 10 mg or matched placebo. The patients are required to take the studied drugs at night (after 21.00 pm) on the first day of chemotherapy and continue daily for six months. Standard treatment is chemotherapy according to each center's standard protocol. Study endpoints are QOL (FACT), adverse event frequency (CTCAE), oxidative stress status, melatonin level, and survival.

ELIGIBILITY:
Inclusion Criteria:

* histologically proven advanced NSCLC, breast, head and neck, sarcoma cancer Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤ 2
* platelet count ≥100,000 cells/mm3
* white blood cell count ≥ 3,000 cell/mm3
* hemoglobin ≥ 10 g/dL
* serum creatinine ≤ 1.5 mg/dL
* bilirubin ≤ 2 mg/dL
* AST ≤ 2.5 times upper limit of normal(ULN)for subjects without metastases or AST ≤ 2.5 times UNL for those with liver metastases
* New York Heart Association grade ≤ 2
* written consent

Exclusion Criteria:

* Patients who receive prior chemotherapy or biotherapy, radiotherapy or surgery within 1 month preceding randomization
* Patients who have more than one type of cancer or brain metastasis were excluded from the trial.
* Patients with moderate neuropathy (CTCAE grade ≥ 2)
* Patients with an active infection, or uncontrolled complications (i.e. blood glucose > 200 mg/dL, uncontrolled hypertension, unstable angina, history of congestive heart failure or history of myocardial infarction within one year).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2007-08; Primary Completion 2011-12 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Quality of Life (FACT) | Change from baseline in total scores at 6 months after treatment
  Self-reported questionnaires. FACT-L, FACT-B, FACT-H&N and FACT-G Thai Version 4 has been previously validated. FACT-L, FACT-B, FACT-H&N and FACT-G are used in lung, breast, head&neck and sarcoma cancer patients, respectively. Change from baseline will be evaluated at 1,2,3 and 6 months after treatment.

SECONDARY OUTCOMES:
Number of participants with adverse events | Baseline and 1,2,3 and 6 months after treatment
  CTCAE Version 4.3
Oxidative stress status | Chemotherapy cycles 1,2,3,4
  8-isoprostane and 8-hydroxydeoxyguanosine urine and MDA plasma analysis
Melatonin level | Chemotherapy cycle 1,2,3 and 4
  Blood, urine and saliva analysis
Overall survival | Over 4 years of the study
  Overall survival

CONTACTS AND LOCATIONS:
Locations (2):
- Thailand (2):
  - Khon Kaen Hospital, Khon Kaen, Changwat Khon Kaen
  - Srinagarind Hospital, Khon Kaen, Changwat Khon Kaen